CLINICAL TRIAL: NCT03752723
Title: A Phase 1b/2, Open Label, Dose Escalation Study to Evaluate Safety, Tolerability, Pharmacodynamics and Antitumor Activity of GX-I7 in Combination With Pembrolizumab in Subjects With Refractory or Relapsed (R/R) TNBC
Brief Title: Study of GX-I7 in Combination With Pembrolizumab in Refractory or Relapsed (R/R) TNBC Subjects(GX-I7-CA-006/KEYNOTE-899)
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Genexine, Inc. (Industry)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: GX-I7-CA-006; KEYNOTE-899 (Other: Merck Sharp & Dohme LLC); MK-3475-899 (Other: Merck Sharp & Dohme LLC)
Record Dates: First submitted 2018-11-19; First posted 2018-11-26 (Actual); Last update posted 2024-03-05 (Actual); Status verified 2024-02

CONDITIONS: Triple Negative Breast Cancer
Keywords: Breast cancer; TNBC
MeSH Terms: conditions — Triple Negative Breast Neoplasms; Breast Neoplasms | interventions — efineptakin alfa; pembrolizumab; Cyclophosphamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- combination with CPA, GX-I7, and pembrolizumab (Experimental): Experimental: combination
  Assigned interventions: CPA, GX-I7 and pembrolizumab
  Interventions: Drug: GX-I7; Drug: Pembrolizumab(KEYTRUDA®); Drug: Cyclophosphamide
- combination with GX-I7, and pembrolizumab (Experimental): Experimental: combination
  Assigned interventions: GX-I7 and pembrolizumab (without CPA)
  Interventions: Drug: GX-I7; Drug: Pembrolizumab(KEYTRUDA®)

INTERVENTIONS:
Drug: GX-I7 — i.m.
  Other Names: Efineptakin alfa
Drug: Pembrolizumab(KEYTRUDA®) — i.v.
  Other Names: KEYTRUDA®; MK-3745
Drug: Cyclophosphamide — i.v.
  Arms: combination with CPA, GX-I7, and pembrolizumab

SUMMARY:
To evaluate the safety and tolerability of escalating doses GX-I7 in combination with standard dose pembrolizumab, and to evaluate objective response rate (ORR) in subjects with refractory or relapsed TNBC

ELIGIBILITY:
Key Inclusion Criteria:

1. Triple negative must be defined as guidelines of American Society of Clinical Oncology(ASCO)/ College of American Pathologist(CAP): Estrogen Receptor (ER) < 1% positive tumor nuclei, Progesterone Receptor (PR) < 1% positive tumor nuclei, and negative for HER2 by IHC 1+, 0 or negativity status confirmed by in situ hybridization (ISH).
2. Subject must have received anthracycline and taxane based chemotherapy for TNBC
3. Has measurable disease as defined by RECIST 1.1 as assessed by the the local site Investigator/radiology.
4. Female subjects, age ≥ 19 years at the time of consent.

Key Exclusion Criteria:

1. Known severe hypersensitivity (≥ Grade 3) to pembrolizumab, pembrolizumab formulation excipients or GX-I7 formulation excipients or cyclophosphamide formulation.
2. Has received prior therapy with an anti-PD-1, anti-PD-L1, or anti-PD-L2 agent or with an agent directed to another co-inhibitory T-cell receptor (ie, CTLA-4, OX-40, CD137) or has previously participated in a Merck pembrolizumab (MK-3475) clinical trial.

Min Age: 19 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 84 (Actual)
Dates: Start 2019-03-27 (Actual); Primary Completion 2023-05-11 (Actual); Study Completion 2023-05-11 (Actual)

PRIMARY OUTCOMES:
Incidence and nature of DLTs | during the first 5 weeks
  To evaluate the safety and tolerability of GX-I7 in combination with standard dose pembrolizumab
Incidence, nature and severity of adverse events | up to 24month
  graded according to NCI CTCAE v5.0
Objective response rate (ORR) | up to 24month
  defined as percentage of subjects with a complete response (CR) or partial response (PR) per RECIST v.1.1

CONTACTS AND LOCATIONS:
Locations (12):
- South Korea (12):
  - Seoul National University Bundang Hospital, Seongnam-si, Gyeonggi-do
  - Ajou Medical Center, Suwon, Gyeonggi-do
  - National Cancer Center, Goyang-si
  - Gachon University Gil Medical Center, Incheon
  - Asan Medical Center, Seoul
  - Ewha Womans University Mokdong Hospital, Seoul
  - Gangnam Severance Hospital, Seoul
  - Korea University Anam Hospital, Seoul
  - Korea University Guro Hospital, Seoul
  - Samsung Medical Center, Seoul
  - Seoul ST.Mary's Hospital, Seoul
  - Severance Hospital, Seoul

IPD SHARING:
Plan to Share IPD: Undecided